CLINICAL TRIAL: NCT02632513
Title: Effect of Passive Ultrasonic Irrigation on Success of Primary Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PGIDS/IEC/2014/120
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Periapical Periodontitis
Keywords: continuous ultrasonic irrigation, syringe irrigation
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous ultrasonic irrigation (Experimental): In continuous ultrasonic irrigation group, Proultra PiezoFlow (Dentsply Tulsa Dental Specialties, Tulsa,OK) was used for the activation of the irrigating solution according to manufacturer's recommendations.
  Interventions: Device: Proultra PiezoFlow (Dentsply Tulsa Dental Specialties)
- Syringe irrigation (No Intervention): In the syringe irrigation group, irrigation was done using 27 gauge syringe.

INTERVENTIONS:
Device: Proultra PiezoFlow (Dentsply Tulsa Dental Specialties) — In continuous ultrasonic irrigation group, Proultra PiezoFlow (Dentsply Tulsa Dental Specialties, Tulsa,OK) was used for the activation of the irrigating solution according to manufacturer's recommendations.
  Arms: continuous ultrasonic irrigation

SUMMARY:
The aim of this study was to compare the success after endodontic treatment performed with or without continuous ultrasonic irrigation.

70 Mandibular molars with diagnosis of pulpal necrosis and with periapical radiolucency were randomly assigned into two treatment groups- continuous ultrasonic irrigation (CUI) and syringe irrigation (SI). Standard nonsurgical endodontic treatment was performed on both groups under rubber dam isolation with 0.02 taper ISO stainless steel hand files using step back technique. In both groups, 5 ml of 5.25% sodium hypochlorite was used as irrigant after each instrument. After root canal instrumentation, canals were irrigated with 5 ml of 17% EDTA solution for 1 minute. In SI group, canals were flushed with 15ml of 5.25% sodium hypochlorite using a 27 gauge needle while final irrigant was delivered using a continuous ultrasonic irrigation device in CUI group. An inter-appointment dressing of calcium hydroxide was given and patient was recalled after one week and canals were obturated with the Gutta Percha. Immediate postoperative radiograph was then taken, followed by radiographs at 3, 6, 9 and 12 months.

DETAILED DESCRIPTION:
Title: Effect of passive ultrasonic irrigation on success of primary endodontic treatment

Introduction:

It is well established that apical periodontitis is caused due to microbial invasion of root canal space. It is an inflammatory disease process comprising host responses to infection of the root canal system of the affected tooth. So, it becomes important to render the root canals free of microorganisms and pathological debris to treat apical periodontitis. Mechanical instrumentation plays an important role in removing microorganisms from the root canal system but it is incapable of rendering canal completely free of bacteria. The intricacies of the root canal system such as fins, isthmi, apical ramifications hinder its complete debridement as these areas are inaccessible to mechanical instrumentation. These complexities continue to harbour bacteria, necrotic tissue and debris and results in persistent periapical inflammation. Thus adjunctive use of root canal irrigant becomes important. Mechanical cleaning of root canals aided by antimicrobial irrigation, thus, are two key elements that help in reducing the bacterial load of root canal and treating apical periodontitis. Irrigation forms an integral part of chemomechanical preparation by facilitating the removal of bacteria, debris and necrotic tissue, especially from areas beyond the reach of root canal instruments. Sodium hypochlorite is recommended as the main irrigant during root canal treatment because of its antimicrobial efficacy as well as its tissue-dissolving capacity but its effectiveness in root canal depends on the irrigant's penetration along the full length of the canal and on irrigant exchange. Although conventional syringe delivery is a well accepted technique of irrigation but it delivers solutions no more than 0-1.1 mm beyond the needle tip thereby limiting irrigant penetration. In addition air entrapment at apical third produces a vapor lock effect, thus impeding the flow of irrigant into the apical region and adequate debridement of the canal system.16 Previous studies have shown that root canals still have detectable levels of cultivable bacteria following chemomechanical procedures with sodium hypochlorite as an irrigant. Consequently, different irrigant agitation techniques have been proposed to increase cleaning efficacy, mechanically and chemically, by enhancing the irrigation dynamics. One such technique is ultrasonic activation of root canal irrigant.

Passive ultrasonic irrigation was first described by Weller et al.The files are designed to oscillate at ultrasonic frequencies of 25-30kHz and operate in a transverse vibration, setting up a characteristic pattern of nodes and antinodes along their length. It enhances irrigant canal wall interaction by transmitting acoustic energy from an oscillating instrument to the irrigant, causing acoustic microstreaming and transient cavitation. Generally for ultrasonic activation of irrigation solution a syringe is used to inject the irrigant into the root canal, after which the irrigant is activated passively by an ultrasonically oscillating instrument. Nascent chlorine, which is the active component responsible for tissue dissolving and antimicrobial action of hypochlorite, is consumed rapidly in such a case. Further, the amount of irrigant that is activated is small, thereby, limiting its debridement efficacy. It has, therefore, been suggested that irrigant delivery methods that provide continuous replenishment of root canal irrigant may be more efficient. Recently, ultrasonic devices have been introduced that provide continuous irrigant delivery along with ultrasonic activation. In these devices irrigating solution moves into the needle through a syringe attached to the luer-lock connection on the needle and is then activated and delivered into the root canal. The main advantages of this technique are the continuous replenishment of the solution and the irrigating solution is delivered from the needle in an activated state, avoiding the need to insert the needle into the apical third of the root canal. Studies have shown that the 1minute of continuous ultrasonic irrigation after hand or rotary instrumentation resulted in significantly cleaner canals and isthmi in the mesial roots of mandibular molars. Carver et al showed that the addition of 1 minute of continuous ultrasonic irrigation significantly reduced bacterial-positive cultures. Another study reported that while continuous ultrasonic irrigation was as effective as intermittent ultrasonic irrigation in the placement of irrigant in the apical part of canal, it led to improved irrigant penetration in lateral canals. In vitro studies comparing continuous ultrasonic irrigation with syringe irrigation in the removal of debris have reported continuous ultrasonic irrigation to be more effective in debris removal from apical third and narrow isthmuses. Curtis et al found that continuous ultrasonic irrigation resulted in significantly less debris present in root canals at 1 and 3 mm from the working length as compared to conventional needle irrigation.A recent study by Layton et al reported that continuous ultrasonic irrigation generates high fluid velocity and shear stress in apical third resulting in enhanced reduction of strictly adherent bacterial biofilm as compared to intermittent ultrasonic irrigation and syringe irrigation.

Whether these parameters translate into better clinical outcome remains to be seen. However, to the best of our knowledge, there is no study assessing the effect of irrigant activation using continuous ultrasonic device on success of endodontic treatment. This randomized controlled trial was therefore designed to evaluate and compare the success of endodontic treatment after the use of continuous ultrasonic irrigation and syringe irrigation.

Methodology: The research project was carried out in the Department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak (Haryana). Protocol of the study was approved by the institutional ethical committee (PGIDS/IEC/2014/120), Rohtak, India and it followed the ethical guidelines of the Helsinki declaration 1975, as revised in 2000. The study was conducted from May 2014 to May 2015.

The study population comprised of patients requiring endodontic treatment following the diagnosis of pulpal necrosis with chronic apical periodontitis in mature mandibular molar. All such patients were examined for establishing their eligibility for the study.

Evaluation of Pulp Vitality Pulp vitality status was evaluated with the help of electric pulp testing, cold testing and clinical evaluation after access opening. If the patient did not respond to electric and thermal test, and no bleeding was observed on access cavity preparation, the subject was included in study provided other inclusion criteria were also met.

Radiographic examination All periapical radiographs were exposed with a 70 kVp machine (Confident, Blue X Imaging S.r.l Via Idiomi 1/8-33 Assago, Italy) using Rinn paralleling device (Dentsply Ltd., Weybridge, Surrey, United Kingdom); and processed manually.

Data gathering Once eligibility was confirmed, the study was explained to the patient and written consent to participate in the study was taken. All the diagnostic, intra operative and post operative findings were recorded on a proforma.

Randomization The patient was randomly assigned to one of the two treatment groups: continuous ultrasonic irrigation (CUI) and syringe irrigation (SI), based on the use of irrigation protocol utilized during chemomechanical preparation. Subjects were assigned to either CUI or syringe irrigation group using an equal proportion allocation ratio. Envelopes that contained concealed assignment codes were assigned sequentially to eligible patients. Both the patient and the operator were blinded of the treatment protocol until completion of chemomechanical preparation.

Clinical Procedure The endodontic treatment was completed in two visits. First Visit Local anaesthesia was administered (2% lidocaine with 1:80000 epinephrine) for patient comfort. The tooth was then isolated with rubber dam. Caries was excavated using round bur in high speed handpiece with copious irrigation and access to the pulp chamber was made. Working length (WL) was obtained with the help of electronic apex locator (Root ZX) using #10 and #15 K file and was confirmed radiographically. The canals were enlarged to a size three sizes larger than the first apical binding file at the working length with 0.02 taper ISO stainless steel hand files, followed by step-back technique with each successively larger file placed 0.5 mm coronal to the previous one. Canal patency was maintained by passing a #10 stainless steel file 0.5 to 1.0 mm beyond the working length. In both the groups, the canals were irrigated with 5 mL of 5.25% sodium hypochlorite (NaOCl) (Hyposol; Prevest Denpro Limited, Jammu, India) solution after every change of instrument using a 27 gauge needle. After shaping, the canals were irrigated with 5 mL 17% EDTA (Prevest Denpro Limited, Jammu, India) for 1 minute.

Post instrumentation irrigation: In continuous ultrasonic irrigation group, Proultra PiezoFlow (Dentsply Tulsa Dental Specialties, Tulsa,OK) was used for the activation of the irrigating solution according to manufacturer's recommendations. The needle was operated using Satelec P5 Piezoelectric Ultrasonic Unit (Acteon, Mount Laurel, NJ) at power setting of 5.The stopper on the PiezoFlow needle was set 1 mm short of binding in the canals, but no more than 75% of the WL. A syringe containing 15 mL of 5.25% NaOCl was attached to the Piezoflow activation needle and the inactive needle was inserted in the canal till premeasured depth, and irrigant flow was started before activation. During activation, the needle was moved up and down passively in the canal, while maintaining the insertion depth to the stopper setting. The irrigation was accomplished in 1 minute per canal at a flow rate of 15 mL/min. In the syringe irrigation group, canals were flushed with 15 ml of 5.25% NaOCl using 27 gauge syringe.

After final irrigation, the canals were dried with sterile absorbent points and filled with calcium hydroxide paste ( Roth International Ltd, Chicago, IL) using a lentulospiral. The tooth was then temporarily restored with Intermediate Restorative Material (Dentsply Ltd, Weybridge, UK).

Second Visit In the second visit, patient returned with completed pain chart and handed it back to the operator. The intracanal dressing was removed with H- files and copious irrigation with 5.25% NaOCl. The master apical Gutta Percha cones were then verified. Canals were obturated with the GuttaPercha and Zinc Oxide- Eugenol based sealer in lateral condensation. After obturation, the access cavity was restored permanently.

An immediate post-operative radiograph was then taken using preset exposure parameters with Rinn paralleling device; and processed manually.

Follow up Follow up clinical and radiographic examination were carried out every 3 months, until 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* • Patient willingness to participate in the study

  * Mature permanent mandibular molar requiring primary root canal treatment
  * Patient's age greater than 18 years
  * There must be radiographic evidence of periapical radiolucency (minimum size ≥ 2.0 × 2.0 mm) and a diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber

Exclusion Criteria:

* • Patients who did not provide authorization for participation in the study

  * Positive history of antibiotic use within past one month of the treatment
  * Positive history of analgesic intake within the past 24 hours
  * Patients who were pregnant, diabetic, immunocompromised, had serious medical illness or required antibiotic premedication
  * Patients with pockets ≥4mm or having marginal of furcal bone loss due to periodontitis
  * Previously accessed teeth and/or with procedural errors
  * Unrestorable tooth, fractured/ perforated roo ts, inflammatory root resorption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Periapical Index score | 1 year
  Change in Periapical Index (PAI) scores (Orstavik et al) observed at 12-months was noted. Scoring of each tooth was done according to the following five point scale (PAI):
  PAI Score Description of radiographic findings
  1. Normal periapical structures
  2. Small changes in bone structure
  3. Changes in bone structure with some mineral loss
  4. Periodontitis with well-defined radiolucent area
  5. Severe periodontitis with exacerbating features

SECONDARY OUTCOMES:
Postoperative pain | 6 hours-7 days
  Visual analog scale (0-100mm) was used to evaluate pain levels. At the end of first appointment, all the patients were instructed to record the level of pain at 6 hours, 12 hours, 18 hours, 24 hours, 2 days, 3 days, 4 days, 5 days, and 6 days on the VAS pain score charts provided after the treatment.